CLINICAL TRIAL: NCT07150897
Title: Early Rehabilitation of Abdominal Muscle Wall Following Lower Transverse Abdominal Incision
Acronym: abdominal reb
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, mohamed naeem, assistant professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMBSUREC/05012025/AWAD; FMBSUREC/05012025/AWAD (Registry Identifier: eman awad); beni suef university (Other: beni suef university)
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: All Participants Are Post Operative Women After Their 1st Cesarean Delivery or Hysterectomy
Keywords: Abdominal Incision, Early Rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study will be designed as a randomized clinical trial that compare 2 groups of participants. Group A (study group) will include participants who join a rehabilitation program starting from day 1 after surgery up to 6 weeks with wearing a belly band. While, group B will involve control participants who follow routine postnatal care as well as wear the same belly band and receive advice as group A participants.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo group (No Intervention): routine postnatal care as well as wear the same belly band and receive advice
- intervention (Experimental): Group A (study group) included participants who join a rehabilitation program starting from day 1 after surgery up to 6 weeks with wearing a belly band
  Interventions: Other: exercise for lower abdominal muscle wall

INTERVENTIONS:
Other: exercise for lower abdominal muscle wall — the exercise session will start with light walking for 5 minutes followed by, posture correction exercises from crock lying, supine, and sitting and standing positions (each exercise will be maintained for 5 seconds and then the woman relaxed for 10 seconds and repeated each exercise 10 times) to overcome the effect of poor pregnancy posture. Then, participants will perform first step of prone plank exercises which is a stable prone plank with attention to maintain a neutral position in the hip joints, pelvis and lumbar spine. The feet will be placed to match the width of the hip and forearm and acted as support points. The elbows place under the glenohumeral joints, and the arms support the body vertically to the surface. Second step of prone plank exercises will involve performing the unilateral stable prone plank which is the same as the stable prone plank but with the dominant leg in a fully extended position. Third step includes, prone bridge on a Swiss Ball with a diameter of 65
  Other Names: Exercise group
  Arms: intervention

SUMMARY:
to investigate effect of inducing rehabilitation program very early after lower abdominal transverse incisions on abdominal muscles.

DETAILED DESCRIPTION:
Abdominal surgery is a general term used to denote surgical procedures conducted in the abdominal area to detect and treat a presenting medical problem.1 Open Abdominal surgery includes vertical and transverse incisions. Low transverse abdominal incision is usually made 1-2 fingerbreadths above the pubic crest with an incision length of 10-14 cm. The lower transverse abdominal incision is adequate for the vast majority of caesarean operations as well as operative disease of the uterus, fallopian tubes, and ovaries. Historically, the gynaecologist- obstetrician has favoured lower abdominal transverse incisions. Several disadvantages of these incisions exist such as limited exploration of the upper abdomen, greater blood loss as well as they are more susceptible to hematoma formation when compared with a midline incision. Paresthesia of the overlying skin results from nerve injury, is more common in a transverse incision compared with a midline incision.2 With regards to the abdominal muscle, there is a relevant surgical related muscle loss induced by major surgical trauma after lower transverse incisions.3 Early postoperative days are associated with fatigue and limited respiratory movements. For the patient, less post operative pain, rapid return to normal function as well as better scar appearance and quality of life are very important factors. Encouraging early mobilization after low transverse abdominal surgery is crucial for optimal healing and recovery of abdominal muscles. In physical therapy, activities such as, transferring from bed to chair, sitting upright, rising from a chair, exercises in or out of bed and walking in the room are considered helpful for surgical patient.4 Up till now, there is no study searched the effect of starting rehabilitation programs for abdominal muscles very early within the first 24 hours after obstetrics and gynaecology surgeries.

ELIGIBILITY:
Inclusion Criteria:a total of 60 women will be recruited from the obstetrics and gynecology Department of Beni-Suef University Hospital, Beni-Suef, Egypt. Their ages will be ranged from 35-50 years and their body mass index (BMI) will not exceed 29 kg/m2. All participants are post operative women after their 1st cesarean delivery or hysterectomy.

-

Exclusion Criteria:Women will be excluded from the study, if they were diagnosed with heart diseases, respiratory diseases causing excessive coughing or sneezing, chronic physical or mental illness, had more than 1 cesarean delivery; had any medical condition that would prohibit active abdominal muscle contraction; or failed to complete an informed consent form.

-

Ages: 35 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-10-17 (Estimated); Study Completion 2025-11-17 (Estimated)

PRIMARY OUTCOMES:
ultrasonography | 4 months
  All assessments will be performed by using a two-dimensional ultrasound diagnostic scanner with a linear probe (Toshiba Xario100, 8-12 MHz linear transducer) to measure thickness of lower part of Rectus Abdominis muscle below umbilicus before and after 6 weeks of the intervention procedure for all participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Beni suef university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
for safty